CLINICAL TRIAL: NCT06428864
Title: Effect of the Use of a 3D Scanner Application on a Smartphone to Mold Garchois Orthotic Device in Neuromuscular Diseases Patients With Scoliosis
Acronym: GSSCAN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0513
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Neuromuscular Diseases; Scoliosis
Keywords: Scoliosis; Neuromuscular Diseases; Orthotic device; Brace; Cast; 3D Scan application
MeSH Terms: conditions — Neuromuscular Diseases; Scoliosis | interventions — Casts, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cast: Patient with a Garchois brace produced after a plaster cast
  Interventions: Device: Plaster cast
- Scan: Patient with a Garchois brace produced after assessment of the thoracic volume with the 3D scan
  Interventions: Device: 3D Scanning

INTERVENTIONS:
Device: Plaster cast — Wearing a Garchois brace produced after a plaster cast
  Groups: Cast
Device: 3D Scanning — Wearing a Garchois brace produced after assessment of the thoracic volume with the 3D scan
  Groups: Scan

SUMMARY:
Neuromuscular scoliosis is the consequence of general hypotonia involved in certain neuromuscular diseases. Thoracic braces are necessary to slow down the deformation. In France, Garchois brace is largely used in this context because of a better pulmonary tolerance.

Historically, molding of thoracic orthotic brace was based on a plaster cast directly on the patient. He/she is suspended in a frame or is lying on an examining table, and is held by 4 therapists (a physician, an orthoprosthesist, a nurse and a doctor). The position during molding could be very uncomfortable and anxious.

With the development of new technologies, a 3D scan application on smartphone to obtain the volume and deformations of the patient was developed. This tool enables digital acquisition of trunk and head volume while bypassing the seated patient. No plaster strips are used. The resulting negative is digitally filled to obtain a positive. The positive is then corrected before the corset is made, either digitally or after 3D scanning, in plaster or foam. This application was first used in our department in 2017.

The aim of this retrospective monocentric study is to show that this application can be used to produce brace that are as corrective and reliable as braces made after plaster casting, while improving the satisfaction of children, their families and professionals during impression taking. as their parents and of the professionals present during the molding.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion or genetically confirmed neuromuscular disease
* Neuromuscular scoliosis, with Garchois brace indication
* Under 18 at the time of the first Garchois brace molding

Exclusion Criteria:

* Other neuro-orthopaedic disease such as cerebral palsy
* Other thoracic brace than Garchois
* Any spine surgery

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Neuromuscular patients from a paediatric rehabilitation center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Cobb angles | Up to 3 months
  Mean differences in Cobb angles measured by spinal X-rays before and after wearing the brace for the 2 groups of patients

CONTACTS AND LOCATIONS:
Locations (1):
- L'Escale - HFME, Bron, France

IPD SHARING:
Plan to Share IPD: No